CLINICAL TRIAL: NCT06062160
Title: The Effect of Therapeutic Touch on Pain and Comfort After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Meltem Akbaş, Assistant Professor, Cukurova University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10.09.2021/114
Record Dates: First submitted 2023-09-20; First posted 2023-10-02 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Therapeutic Touch; Postpartum Period; Midwifery; Comfort
Keywords: Therapeutic Touch; comfort; midwifery; pain; postpartum period
MeSH Terms: conditions — Pain | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: There is a difference between the posttest pain scores of the intervention group and the control group.
  There is a difference between the comfort level posttest scores of the intervention group and the control group.
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental group received deep Therapeutic Touch two time at 10th and 40nd hours after cesarean section.
  Interventions: Other: Therapeutic Touch
- Control (No Intervention): There will be no intervention in the control group. Routine maintenance will be given.

INTERVENTIONS:
Other: Therapeutic Touch — Experimental group received deep Therapeutic Touch two time at 10th and 40nd hours after cesarean section.
  Arms: Experimental

SUMMARY:
This study was conducted as randomized controlled study to evaluate the effect of Therapeutic Touch on acute pain and comfort level in women who delivered by cesarean section. Personal information form was used as data collection form, VAS was used to assess pain, and PPCQ was used to assess comfort. When power analysis was performed, the sample size was calculated to be at least 45 participants for each group (45 experiments, 45 controls). Experimental group received deep Therapeutic Touch by investigators two time at 10th and 40nd hours after cesarean section.

DETAILED DESCRIPTION:
Cesarean section rate is increasing in the world and in our country, and it might bring other problems with it. Pain, breastfeeding problems and decrease in comfort problems have high chance to happen after cesarean section. The insufficiency of pharmacological methods in reducing the problems experienced after cesarean section and having many side effects increase the using percentage tendency to non-pharmacological methods.

This study was conducted as randomized controlled study to evaluate the effect of Therapeutic Touch on acute pain and comfort level in women who delivered by cesarean section. Personal information form was used as data collection form, VAS was used to assess pain, and PPCQ was used to assess comfort. When power analysis was performed, the sample size was calculated to be at least 45 participants for each group (45 experiments, 45 controls). Experimental group received deep Therapeutic Touch by investigators two time at 10th and 40nd hours after cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* • Those between the ages of 18 and 45

  * Multiparous women
  * At the 8th postoperative hour
  * Women who have not developed any complications during pregnancy, birth and postpartum for themselves or their newborns.
  * Having a single, healthy newborn at term,
  * Does not react negatively to any attempt to touch,
  * Able to speak and communicate in Turkish
  * Agreeing to participate in the study

Exclusion Criteria:

* Those with any problems diagnosed before or at birth (such as oligohydramnios, preeclampsia, heart disease, diabetes, placenta previa)
* Those who develop any complications related to mother and baby in the postpartum period (bleeding, hypertension, babies taken to the neonatal intensive care unit, etc.).
* Those who receive different analgesics other than routine post-operative analgesics (75 mg diclofenac sodium in the first 30 minutes post-op).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Measurement was taken half an hour after the intervention.
  The scale is scored between 0-10 points. As the score increases, the pain increases.
Postpartum Comfort Scale | Measurement was taken half an hour after the intervention.
  The scale is scored between 34 and 170 points. As the score increases, comfort increases.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Akbaş, PhD, Principal Investigator — Universty Of Cukurova
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No